CLINICAL TRIAL: NCT02281357
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Tralokinumab in Reducing Oral Corticosteroid Use in Adults and Adolescents With Oral Corticosteroid Dependent Asthma (TROPOS)
Brief Title: Phase 3 Study to Evaluate the Efficacy & Safety of Tralokinumab in Adults & Adolescents With OCS Dependent Asthma
Acronym: TROPOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2210C00013
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-02

CONDITIONS: Asthma
Keywords: Asthma; Reactive Airways; Repiratory Tract Disease; Obstructive Lung Disease; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases, Obstructive; Lung Diseases | interventions — tralokinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralokinumab (Experimental): Tralokinumab subcutaneous injection
  Interventions: Biological: Tralokinumab
- Placebo (Placebo Comparator): Placebo subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tralokinumab — Tralokinumab dose
  Arms: Tralokinumab
Other: Placebo — Placebo dose
  Arms: Placebo

SUMMARY:
A Multicentre, Randomized, Double-blind, Parallel Group, Placebo Controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Tralokinumab in Reducing Oral Corticosteroid dependent Asthma.

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel group, placebo-controlled study designed to evaluate the efficacy and safety of a fixed 300 mg dose of tralokinumab administered subcutaneously every 2 weeks in adult and adolescent subjects with oral corticosteroid dependent asthma. Approximately120 subjects will be randomized globally. Subjects will receive tralokinumab or placebo, administered via subcutaneous injection at the study site, over a 40-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

1) Age 12-75 2) Documented physician-diagnosed asthma. 3) Documented treatment with ICS at a total daily dose corresponding to ≥500µg fluticasone propionate dry powder formulation and a LABA. 4) Subjects must have received OCS for the treatment of asthma for 6 months prior to Visit 1 and on a stable OCS dose between ≥7.5 to ≤30mg daily or daily equivalent for at least one month prior to enrolment (Visit 1) . 5) Pre-BD FEV1 value <80% (<90% for patients 12-17 yrs of age) of their PNV. 6) Post-BD reversibility of ≥12% in FEV1.

Exclusion Criteria:

1) Clinically important pulmonary disease other than asthma. 2) History of anaphylaxis following any biologic therapy. 3) Hepatitis B, C or HIV. 4) Pregnant or breastfeeding. 5) History of cancer. 6) Current tobacco smoking or a history of tobacco smoking for ≥10 pack-years. 7) Previous receipt of tralokinumab.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2017-09-07 (Actual); Study Completion 2017-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William W Busse, M.D., Principal Investigator — University of Wisconsin School of Medicine and Public Health, Department of Medicine, Allergy & Immunology
Locations (46):
- United States (15):
  - Research Site, New Haven, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, St Louis, Missouri
  - Research Site, Rochester, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Monroeville, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Tyler, Texas
  - Research Site, Richmond, Virginia
- Belgium (5):
  - Research Site, Brussels (Anderlecht)
  - Research Site, Ghent
  - Research Site, Hasselt
  - Research Site, Leuven
  - Research Site, Woluwé-St-Lambert
- France (5):
  - Research Site, Grenoble
  - Research Site, Lille
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Pessac
- Germany (7):
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mainz
  - Research Site, München
  - Research Site, München-Pasing
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Leeuwarden
- Poland (7):
  - Research Site, Bystra
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Rzeszów
  - Research Site, Wroclaw
- Ukraine (4):
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Vinnytsia

REFERENCES:
- [Background] Busse WW, Brusselle GG, Korn S, Kuna P, Magnan A, Cohen D, Bowen K, Piechowiak T, Wang MM, Colice G. Tralokinumab did not demonstrate oral corticosteroid-sparing effects in severe asthma. Eur Respir J. 2019 Jan 31;53(2):1800948. doi: 10.1183/13993003.00948-2018. Print 2019 Feb. PMID 30442714
- [Derived] Panettieri RA Jr, Wang M, Braddock M, Bowen K, Colice G. Tralokinumab for the treatment of severe, uncontrolled asthma: the ATMOSPHERE clinical development program. Immunotherapy. 2018 Mar 1;10(6):473-490. doi: 10.2217/imt-2017-0191. Epub 2018 Mar 14. PMID 29536781
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2966&filename=d2210c00013-revised-csp-4_Redacted_PDFA.pdf
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=2966&filename=d2210c00013-sap-ed-3_redaction_proposed_Redacted_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 19 February 2015; Last patient last visit: 07 September 2017. Study performed at 56 sites in 7 countries. Patients were maintained on their currently prescribed inhaled corticosteroid long-acting β2-agonist therapy and any additional asthma controller medications throughout the study period.
Pre-assignment Details: 218 patients were screened. Prior to randomisation, patients completed a run-in period or run-in/oral corticosteroid (OCS) optimisation period (reached their minimum effective dose of OCS and remained stable on that dose for 2 weeks). 140 patients were randomised to study treatment. All randomised patients received study treatment.
Groups:
- Tralokinumab: Tralokinumab 300 milligrams (mg) administered by subcutaneous (SC) injection every two weeks (Q2W) over a 40-week treatment period.
- Placebo: Placebo was administered by SC injection over a 40-week treatment period.
Period: Overall Study
Arm/Group | Tralokinumab | Placebo
Started | 70 | 70
Completed (Patients who completed treatment and patients who discontinued treatment but completed the study.) | 63 | 66
Not Completed | 7 | 4
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 4 | 3

BASELINE CHARACTERISTICS:
Population: All patients in the full analysis set (FAS) who received any study treatment (tralokinumab or placebo) were included in the baseline analysis.
Groups:
- Tralokinumab: Tralokinumab 300 mg administered by SC injection Q2W over a 40-week treatment period.
- Total: Total of all reporting groups
Arm/Group | Tralokinumab | Placebo | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 58 | 55 | 113
  >=65 years | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.05) | 55.4 (10.26) | 54.7 (10.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 39 | 87
  Male | 22 | 31 | 53
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 66 | 63 | 129
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Final Daily, Average, OCS Dose at Week 40 While Not Losing Asthma Control.
Description: The 40-week treatment period consisted of 3 phases: an induction phase (Week 0 to Week 12) where patients remained on their optimised OCS dose; an OCS reduction phase (Week 12 to Week 32) where OCS dose reduction could have started at Week 12 with the possibility of dose titration every 4 weeks to reach the lowest possible OCS dose; and a maintenance phase (Week 32 to Week 40) where patients remained on the OCS dose reached at Week 32 to demonstrate asthma control was maintained after achieving the lowest OCS dose. Criteria used to assess asthma control included lung function assessments (forced expiratory volume in 1 second and morning peak expiratory flow), night awakenings, and the use of rescue medication and systemic corticosteroids.
  The least squares (LS) mean percent change from baseline in average daily OCS dose is presented. The final daily percent change from baseline was defined as {(Final daily average dose - baseline daily average dose)/baseline daily average dose}*100%.
Time Frame: Baseline (Week 0) and Week 40
Population: The FAS included all randomised patients who received at least one dose of study treatment, irrespective of their protocol adherence and continued participation in the study.
Measure: Least Squares Mean (Standard Error); unit: Percent change from baseline
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 70 | 70
Percent change from baseline | -37.62 (4.98) | -29.85 (4.98)
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Comparison of percent change from baseline in OCS dose: tralokinumab vs placebo; Test type: Superiority — The null hypothesis was that the average percentage change in OCS dose on tralokinumab was equal to the average percentage change in OCS dose on placebo; p = 0.271, ANCOVA; The analysis of covariance (ANCOVA) model utilised a sandwich estimator for the variance; LS Mean difference = -7.78, 95% CI 2-sided [-21.70 to 6.15] — The model included treatment group as a fixed effect and baseline OCS dose as a continuous covariate. No interaction terms were included in the model. All group comparisons from the ANCOVA model were based on Type III sums of squares

2. Secondary Outcome: The Number of Patients With Final Daily Average OCS Dose ≤5 mg at Week 40.
Description: The 40-week treatment period consisted of 3 phases: an induction phase (Week 0 to Week 12) where patients remained on their optimised OCS dose; an OCS reduction phase (Week 12 to Week 32) where OCS dose reduction could have started at Week 12 with the possibility of dose titration every 4 weeks to reach the lowest possible OCS dose; and a maintenance phase (Week 32 to Week 40) where patients remained on the OCS dose reached at Week 32 to demonstrate asthma control was maintained after achieving the lowest OCS dose.
  The number of patients with a final daily average OCS dose ≤5.0 mg is presented. For patients prescribed a fixed daily dose, then the average OCS dose was defined as the prescribed dose. For patients on a regimen where a different amount of OCS was to be taken each day, then the average OCS dose was defined as the average amount prescribed to be taken each day.
Time Frame: At Week 40
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 70 | 70
Participants | 32 | 28
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Comparison of OCS dose ≤5.0 mg: tralokinumab vs placebo; Test type: Superiority; p = 0.442, Regression, Logistic; The model included treatment group as a fixed effect and baseline OCS dose as a continuous covariate; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.65 to 2.73]

3. Secondary Outcome: The Number of Patients With ≥50% Reduction in Final Average Daily OCS Dose at Week 40.
Description: The 40-week treatment period consisted of 3 phases: an induction phase (Week 0 to Week 12) where patients remained on their optimised OCS dose; an OCS reduction phase (Week 12 to Week 32) where OCS dose reduction could have started at Week 12 with the possibility of dose titration every 4 weeks to reach the lowest possible OCS dose; and a maintenance phase (Week 32 to Week 40) where patients remained on the OCS dose reached at Week 32 to demonstrate asthma control was maintained after achieving the lowest OCS dose.
  The number of patients with ≥50% reduction in average daily OCS dose is presented. The final daily percent change from baseline was defined as {(Final daily average dose - baseline daily average dose)/baseline daily average dose}*100%. If this resulted in a value of -50% or less (more negative), that patient was classified as having at least a 50% reduction in final daily average OCS dose.
Time Frame: At Week 40
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 70 | 70
Participants | 31 | 26
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Comparison of ≥50% reduction in OCS dose: tralokinumab vs placebo; Test type: Superiority; p = 0.356, Regression, Logistic; The model included treatment group as a fixed effect and baseline OCS dose as a continuous covariate; Odds Ratio (OR) = 1.38, 95% CI 2-sided [0.70 to 2.74]

4. Secondary Outcome: Annual Asthma Exacerbation Rate (AAER) up to Week 40.
Description: AAER up to Week 40 in the tralokinumab group was compared to that seen in the placebo group. The response variable was the number of exacerbations the patient experienced up to Week 40, with the logarithm of the time at risk in years of experiencing an exacerbation included as offset in the model.
  AAER = number of exacerbations*365.25/(follow-up date - date of randomisation + 1).
  Asthma exacerbation was defined as a worsening of asthma that led to any of the following:
  * Use of systemic corticosteroids for at least 3 days; a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of systemic corticosteroids.
  * An emergency room (ER) or urgent care (UC) visit (defined as evaluation and treatment for <24 hours in an ER or UC centre) due to asthma that required systemic corticosteroids.
  * An inpatient hospitalisation (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma.
Time Frame: Baseline (Week 0) up to Week 40
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Adjusted rate (events/year)
Arm/Group | Tralokinumab | Placebo
Number analyzed (Participants) | 70 | 70
Adjusted rate (events/year) | 1.84 [1.43 to 2.36] | 2.31 [1.83 to 2.92]
Statistical Analysis 1: Comparison: Tralokinumab vs Placebo; Comparison of AAER: tralokinumab vs placebo; Test type: Superiority; p = 0.186, Negative binomial; Rate Ratio = 0.80, 95% CI 2-sided [0.57 to 1.12] — Treatment group, OCS dose at baseline, and number of exacerbations in the previous year are included in the model as covariates

ADVERSE EVENTS:
Time Frame: 40 weeks.
Description: Data is reported for adverse events with an onset date ≥ the first day of study treatment and ≤ (the last day of study treatment + 2 weeks). Patient population was the safety analysis set which included all patients who received at least one dose of study treatment.
Groups:
- Tralo 300 mg Q2W: Tralokinumab 300 mg administered by SC injection Q2W over a 40-week treatment period.
Arm/Group | Tralo 300 mg Q2W | Placebo
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70
Serious Adverse Events (participants affected / at risk) | 9/70 | 16/70
Other Adverse Events (participants affected / at risk) | 55/70 | 44/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=70) | Placebo (N=70)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary function test abnormal (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 8 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tralo 300 mg Q2W (N=70) | Placebo (N=70)
Fatigue (General disorders) | 3 (3) | 5 (6)
Injection site erythema (General disorders) | 6 (13) | 0 (0)
Injection site pain (General disorders) | 6 (12) | 2 (2)
Injection site pruritus (General disorders) | 5 (6) | 0 (0)
Bronchitis (Infections and infestations) | 11 (12) | 16 (20)
Oral candidiasis (Infections and infestations) | 2 (2) | 4 (4)
Sinusitis (Infections and infestations) | 5 (7) | 4 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Viral upper respiratory tract infection (Infections and infestations) | 25 (33) | 10 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Headache (Nervous system disorders) | 14 (33) | 11 (15)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-02-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT02281357/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT02281357/SAP_001.pdf